CLINICAL TRIAL: NCT06271876
Title: Influence of an Inspiratory Muscle Fatigue Protocol on Healthy Youngs on Respiratory Muscle Strength, Vertical Jump Performance and Muscle Oxygen Saturation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sierra Varona SL (Other)
Collaborators: Universidad Europea de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0011
Record Dates: First submitted 2024-02-12; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: the outcome assessor will not know in which group is each participant, and the investigator will receive the data without knowing which data is from which group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Inspiratory muscle fatigue group (Experimental): The EG (experimental group) will perform the diaphragmatic fatigue protocol using a specific inspiratory endurance test, in which volunteers, one-on-one, and in a single session, will breathe against submaximal inspiratory loads equivalent to 60% of their MIP (Maximum Inspiratory Pressure) through a threshold valve device. The participants will follow a free pattern of breathing until they are unable to establish flow during at least 3 maximum inspiratory efforts.
  Interventions: Other: Inspiratory muscle training
- Control group (No Intervention): they will not receive any intervention. Just sit and wait the same amount of time that the intervention and the activation group needs to finish their protocol (around 10 minutes)
- Inspiratory muscle activation group (Active Comparator): The activation group will perform the protocol of 2 sets of 30 repetitions at 40% of their MIP, one-on-one, and in a single session, breathing against submaximal inspiratory loads using a threshold valve device. The participants will follow a free pattern of breathing until complete the protocol.
  Interventions: Other: Inspiratory muscle training

INTERVENTIONS:
Other: Inspiratory muscle training — The subjects will perform deep inspirations against a threshold device with varying resistances
  Other Names: Inspiratory muscle fatigue
  Arms: Inspiratory muscle activation group; Inspiratory muscle fatigue group

SUMMARY:
Respiratory muscle training represents an effective method increasingly utilized in both sports and healthcare domains, employing various devices, among which threshold devices are prominent. The aim of this study is to determine the relationship between inspiratory muscle fatigue and muscular strength in lower limbs, in both healthy and pathological subjects, as well as the association between such fatigue and other variables, including maximal inspiratory pressure and muscle tissue oxygen levels.

According to our hypothesis, the execution of a protocol inducing inspiratory muscle fatigue in healthy youngs could influence muscular strength, exercise capacity and muscle tissue oxygenation.

In this study, subjects will be divided into three groups: experimental group , activation group and control group.

Measurements of variables, such as maximal inspiratory pressure, peripheral muscle tissue oxygen levels, diaphragmatic strength (ultrasound image) and vertical jump performance, will be conducted.

DETAILED DESCRIPTION:
This is a randomized control trial. Experimental group (EG) will perform an inspiratory muscle fatigue protocol using a specific inspiratory endurance test, in which volunteers, one-on-one, and in a single session, will breathe against submaximal inspiratory loads equivalent to 60% of their Maximum Inspiratory Pressure (MIP) through a threshold valve device. Participants will follow a free pattern of breathing until they are unable to establish flow during at least 3 maximum inspiratory efforts.

Activation group (AG) will perform a protocol of 2 sets of 30 repetitions at 40% of their MIP, one-on-one, and in a single session, using a threshold valve device.

Control group will do a seat and wait.

Interventions will be supervised by a physiotherapist. Primary outcomes will be:

Muscle oxygen saturation (SmO2) will be assessed using a near infrared spectroscopy device, immediately before intervention and immediately after intervention.

Vertical jump performance will be assessed by Counter Movement Jump (CMJ) test. CMJ test involved starting from a standing position with hands placed on hips, followed by a rapid upward jump achieved by flexing and extending knees. This plyometric action followed sequence of "eccentric - isometric - concentric" movements. CMJ measurements were taken using a force platform. This will be done immediately before intervention and immediately after intervention

Respiratory muscle strength will be assessed using a respiratory pressure meter or manometer designed, and with ultrasound image measuring cross sectional area of diaphragm at 8-9th rib level and speed of contraction with a deep and fast inspiratory manoeuver. This will be done immediately before intervention and immediately after intervention

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-45 years.
* Non-smoker.
* Engaged in sports activity at least 3 times a week for a minimum of one year.

Exclusion Criteria:

* Having a medical condition that impedes engaging in physical activity.
* Individuals with compromised cognitive capacities.
* Subjects with any chronic disease (cardiorespiratory, neurological, metabolic, oncological, etc.).
* Subjects with tympanic perforation or middle-inner ear pathology.
* Subjects who have undergone lower limb surgery within the past 12 months.
* Subjects experiencing an active episode of lower limb pain.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-03-03 (Estimated); Primary Completion 2024-03-09 (Estimated); Study Completion 2024-03-19 (Estimated)

PRIMARY OUTCOMES:
Respiratory muscle strength | Pre intervention and immediately post intervention
  It will be assessed using a MicroRPM® (MicroMedical, UK).The MicroRPM® is likely a respiratory pressure meter or manometer designed for measuring respiratory muscle strength. It typically includes a mouthpiece connected to a pressure sensor, and the device measures the force or pressure generated during respiratory maneuvers.
  The person will be instructed to take a maximal deep breath in, and then exhale to residual volume. After that, they will be asked to inhale forcefully against the resistance provided by the MicroRPM®. This measures the strength of the inspiratory muscles.
  The measures will be expressed in cmH2O.
Diaphragmatic thickness and thickening fraction | Pre intervention and immediately post intervention
  Diaphragmatic thickness and thickening fraction The linear array probe with a frequency of 3.0-10 megahertz (MHz) is placed perpendicularly to chest wall close to the mid-axillary line which is between the 8th and 10th intercostal space. The thickness of diaphragm is measured at the end of expiration and maximum inspiration for three times and the average values were recorded.
  The measures will be expressed in centimeters.
Diaphragm movement curve | Pre intervention and immediately post intervention
  The convex array probe with a frequency of 1.5-4.6 MHz is placed below the midclavicular line of the right costal margin in longitudinal scanning plane. The liver was used as an inspection window, and the probe was pointed toward the cephalic side. The ultrasound bundle is perpendicular to the posterior third of the right diaphragm. M-mode ultrasound is used to record the diaphragmatic movement curve during quiet breathing (QB) and deep breathing (DB).
  The measures will be expressed in seconds.
Vertical jump performance | Pre intervention and immediately post intervention
  The Counter Movement Jump (CMJ) test involved starting from a standing position with hands placed on the hips, followed by a rapid upward jump achieved by flexing and extending the knees. This plyometric action followed the sequence of "eccentric - isometric - concentric" movements. The CMJ measurements were taken using the force platform

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Ladriñán Maestro, Principal Investigator — Universidad Europea de Madrid

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ladrinan-Maestro A, Sanchez-Infante J, Martin-Vera D, Sanchez-Sierra A. Influence of an inspiratory muscle fatigue protocol on healthy youths on respiratory muscle strength, vertical jump performance and muscle oxygen saturation: a randomized controlled trial. J Transl Med. 2024 Aug 5;22(1):732. doi: 10.1186/s12967-024-05555-3. PMID 39103816